CLINICAL TRIAL: NCT02139774
Title: Feasibility of an Evidence-based Walking Program in a Sample of Men Age >65 Undergoing Treatment for Prostate Cancer
Brief Title: Using Walk With Ease Walking Program With Men 65 and Older Being Treated for Prostate Cancer
Status: Terminated | Type: Observational
Why Stopped: inadequate accrual
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1320; 13-2929 (Other: UNC IRB)
Record Dates: First submitted 2014-02-26; First posted 2014-05-15 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Elderly; Geriatric; Radiation; Arthritis; Exercise; Walking; Endocrine Therapy; Androgen Deprivation Therapy; Active Surveillance; Men
MeSH Terms: conditions — Prostatic Neoplasms; Arthritis; Motor Activity; Multiple Endocrine Neoplasia Type 1 | interventions — Walking; methyl hydroxyethyl cellulose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Active Survelliance: Men age 65 and older who are undergoing active surveillance as primary treatment for their prostate cancer.
  Interventions: Behavioral: Walk with Ease
- Radiation: Men age 65 and older who are undergoing radiation only as primary treatment for their prostate cancer.
  Interventions: Behavioral: Walk with Ease
- Endocrine Therapy: Men age 65 and older who are undergoing endocrine therapy as primary treatment for their prostate cancer.
  Interventions: Behavioral: Walk with Ease
- Surgery: Men age 65 and older who are undergoing surgery as primary treatment for their prostate cancer.
  Interventions: Behavioral: Walk with Ease

INTERVENTIONS:
Behavioral: Walk with Ease — A six week walking program by the Arthritis Foundation

SUMMARY:
This study is testing a walking program called Walk with Ease by the Arthritis Foundation with men undergoing treatment for prostate cancer. The researchers are interested in how easy or difficult it is for these men to participate in this program and whether or not is is helpful to them during their care.

DETAILED DESCRIPTION:
Purpose: This pilot study evaluates the feasibility of implementing a moderate-intensity physical activity (PA) program in a sample of men age 65 or older with a prostate cancer diagnosis undergoing various forms of treatment or active surveillance.

Participants: Men, 65 and older, with a prostate cancer diagnosis.

Procedures (methods): This study will enroll subjects in a 6 week walking program called Walk with Ease (WWE) and see if walking can be sustained for up to three months. In addition, the study will perform a Geriatric Assessment and gather preliminary data on self-reported quality of life outcomes and self-reported physical activity as captured in a daily walking log.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years of age
* Histologically confirmed Stage I, II or III prostate cancer (endocrine (± radiation) patients may be Stage IV)
* Undergoing prostate cancer treatment (post-surgery only, radiation only, endocrine therapy (± radiation), or active surveillance)
* English speaking
* IRB approved, signed written informed consent
* Approval from their treating physician to engage in moderate-intensity physical activity
* Patient-assessed ability to walk and engage in moderate physical activity
* Willing and able to meet all study requirements

Exclusion Criteria:

* One or more significant medical conditions that in the physician's judgment preclude participation in the walking intervention
* Major surgery scheduled within the study period
* Unable to walk or engage in moderate-intensity physical activity
* Already actively walking (150 minutes per week)

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Men aged 65 and older with Prostate Cancer
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To measure the feasibility of implementing the WWE intervention among men age >65 with a prostate cancer diagnosis | 24 months
  Exploring the evaluate the feasibility of implementing the WWE intervention among men age >65 with a prostate cancer diagnosis. The study will measure those who were able to complete the program and increased their self-reported level of walking. The study will also measure the percent of patients who reach the goal of walking 30 minutes a day for 5 days a week in order to determine feasibility.

SECONDARY OUTCOMES:
Measure the rate of completion for study surveys | 24 months
  To evaluate the rate of completion of each of the following measures/assessments at 3 different time points -- baseline, 6 weeks (end of WWE intervention), and 3 months (follow-up):
  * Self-reported walking log
  * Functional Assessment of Cancer Therapy-General (FACT-G)25
  * Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue26
  * Outcome Expectations for Exercise (OEE) scale27
  * Perceived Self-Efficacy for Fatigue Self-Management (PSEFSM)28,29
  * Visual Analog Scales (VAS) for Pain, Fatigue and Stiffness30-32
  * PROMIS Pain Interference Short Form 6b33-35
  * BRFSS Questionnaire 2011 -Health Behaviors Questionnaire (HBQ)36
  * Geriatric Assessment (GA) (Version 5)

OTHER OUTCOMES:
Use primary data to design future studies | 36 months
  To explore data from the measures/assessments (summary measures at each time point and mean changes at 6 weeks and 3 months) to inform future studies designed to evaluate associations between the WWE program and these variables.

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Muss, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Website for the Geriatric Oncology program at UNC Chapel Hill — http://unclineberger.org/geriatric